CLINICAL TRIAL: NCT01332591
Title: Multivessel Coronary Disease Diagnosed at the Time of Primary PCI for STEMI: Complete Revascularization Versus Conservative Strategy. PRAGUE - 13 Trial
Brief Title: Multivessel Disease Diagnosed at the Time of PPCI for STEMI: Complete Revascularization Versus Conservative Strategy.
Acronym: Prague-13
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Anne's University Hospital Brno, Czech Republic (Other)
Collaborators: Bulgarian Cardiac Institute (Network); Tomas Bata Hospital, Czech Republic (Other)
Responsible Party: Principal Investigator, Ota Hlinomaz, MD, PhD, Ota Hlinomaz, MD, PhD, St. Anne's University Hospital Brno, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NT11412
Record Dates: First submitted 2011-03-30; First posted 2011-04-11 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Coronary Artery Stenosis
Keywords: STEMI, primary PCI, non-infarct, non-culprit lesion, CABG
MeSH Terms: conditions — Coronary Stenosis; ST Elevation Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Complete revascularization (Active Comparator): Percutaneous coronary intervention of "non-infarct" coronary arteries
  Interventions: Procedure: Percutaneous coronary intervention
- Conservative management (No Intervention): standard guideline-based medical therapy

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — PCI of significant stenoses of "non-infarct" coronary arteries
  Arms: Complete revascularization

SUMMARY:
The aim of the study is to find the optimal management of patients with acute myocardial infarction with ST elevations treated by primary PCI who have at least one significant stenosis of non-culprit coronary artery. The primary endpoint of the study will be incidence of combined endpoint of all cause mortality, nonfatal myocardial infarction and stroke during the follow up of 24 months in group of patients treated with staged revascularization (PCI or CABG) in comparison with patients treated conservatively.

DETAILED DESCRIPTION:
Introduction:

Primary percutaneous coronary intervention (PPCI) of the occlussion or significant stenosis of infarct artery is a method of choice in treatment of acute myocardial infarction with ST segment elevation (STEMI). It is not clear, what is the optimal management of patients with acute myocardial infarction with ST elevations (STEMI) treated by primary percutaneous coronary intervention (PPCI) who have at least one significant stenosis of non-culprit coronary artery. Numerous cardiology centers perform staged PCI on significant stenoses involving the "non-infarct" coronary artery (arteries) 3-40 days after PPCI, but the benefit of this staged PCI for such patients has not yet been clearly demonstrated.

Aim of study:

The aim is to find the optimal management of patients with acute myocardial infarction with ST elevations (STEMI) treated by PPCI who have at least one significant stenosis of non-culprit coronary artery. The primary endpoint of the study will be incidence of combined endpoint of all cause mortality, nonfatal myocardial infarction and stroke during the follow up of 24 months in group of patients treated with staged revascularization (PCI or CABG) in comparison with patients treated conservatively.

Hypothesis:

Our hypothesis is that complete staged revascularization of significant stenoses of the coronary arteries will improve the long-term prognosis in patients after PPCI as compared to conservative management.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acute myocardial infarction with ST segment elevation (STEMI)
* Angiographically successful primary PCI of infarct-related stenosis (TIMI flow grades II-III)
* One or more other stenoses (≥70%) of "non-infarct" coronary artery (arteries) found by coronary angiography, (diameter of artery ≥ 2,5mm)
* Enrollment ≥48 hours following onset of symptoms

Exclusion Criteria:

* Stenosis of the left main of left coronary artery ≥ 50%
* Hemodynamically significant valvular disease
* Patients in cardiogenic shock during STEMI
* Hemodynamic instability
* Angina pectoris > grade 2 CCS lasting 1 month prior to STEMI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2008-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
composite endpoint of death, nonfatal acute myocardial infarction and stroke | 2 years

SECONDARY OUTCOMES:
cardiovascular death | 2 years
recurrent myocardial infarction | 2 years
target vessel failure | 2 years
  progression of studied stenosis of non-culprit artery
stroke | 2 years
hospitalization for heart failure | 2 years
changes of left ventricular ejection fraction | 2 years
hospitalization for unstable angina pectoris | 2 years
outcomes of questionnaire regarding angina pectoris | 2 years
target vessel revascularization | 2 years
  non infarct artery
target lesion revascularization | 2 years
  non infarct artery

CONTACTS AND LOCATIONS:
Overall Officials: Ota Hlinomaz, MD, PhD, Principal Investigator — +420604273627
Locations (1):
- Department of Cardioangiology, St. Anne University Hospital, Brno, Czechia